CLINICAL TRIAL: NCT00197210
Title: A Phase III, Double-blind, Randomized, Placebo-controlled, Multi-country and Multi-center Study to Assess the Efficacy and Safety of Two Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine in Healthy Infants
Brief Title: A Study to Test 2 Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 444563/028/029/030; 444563/029 (Other: GSK); 444563/030 (Other: GSK)
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Infections, Rotavirus
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Biological: Rotavirus

SUMMARY:
The main objectives of this study are to determine vaccine efficacy against severe rotavirus (RV) gastroenteritis (GE) during the period starting from 2 weeks after Dose 2 until two years of age and to determine the safety of GSK Biologicals' HRV vaccine with respect to definite intussusception (IS) within 31 days (Day 0-Day 30) after each HRV vaccine dose.

DETAILED DESCRIPTION:
The study has two groups: Group HRV and Group Placebo. Two oral doses administered to healthy infants who are 6-12 weeks of age in Hongkong and Taiwan or 11-17 weeks of age in Singapore, according to a 0, 1 to 2-month schedule. Routine vaccinations are given concomitantly with the study vaccines at 2 or 3 and 4 months of age according to each local country regulation. Whenever OPV is used, a minimum 2-week interval should be observed between HRV vaccine and OPV doses.

ELIGIBILITY:
Inclusion criteria:

* Healthy infants 6-12 or 11-17 weeks of age at the time of dose 1 whose parent/guardian sign a written informed consent and whose parents/guardians can and will comply with the requirements of the protocol.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine or placebo, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Child is unlikely to remain in the study area during study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine.
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period.
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal tract or other serious medical condition as determined by the investigator.
* First or second degree of consanguinity of parents.

Ages: 6 Weeks to 17 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10708 (Actual)
Dates: Start 2003-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of severe RV GE caused by the wild RV strains from 2 weeks after Dose 2 until two years of age. Occurrence of definite IS cases within 31 days (Day 0 -Day 30) after each HRV vaccination dose.

SECONDARY OUTCOMES:
Severe RV GE by wild-type G1, non-G1, each non-G1 and severe GE from 2 weeks after Dose 1 and 2 until 2-year old. SAEs. Mortality. Definite IS until 2-years old. Serum anti-RV IgA at Visits 1 and 3 (100 subjects/country).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Guillermo M et al. RIX4414 (Rotarix™) has demonstrated efficacy during the first 2 years of life in infants from 11 Latin American countries. Abstract presented at the 10th International Rotavirus Symposium (IRS), Bangkok, Thailand, 19-21 Sep 2012.
- [Background] Lau YL, Nelson EA, Poon KH, Chan PK, Chiu S, Sung R, Leung CW, Ng D, Ma YM, Chan D, Lee TL, Tang J, Kwan YW, Ip P, Ho M, Fung LW, Tang H, Suryakiran PV, Han HH, Bock H; Hong Kong Rotarix Study Group. Efficacy, safety and immunogenicity of a human rotavirus vaccine (RIX4414) in Hong Kong children up to three years of age: a randomized, controlled trial. Vaccine. 2013 Apr 26;31(18):2253-9. doi: 10.1016/j.vaccine.2013.03.001. Epub 2013 Mar 13. PMID 23499605
- [Background] Phua KB, Lim FS, Lau YL, Nelson EA, Huang LM, Quak SH, Lee BW, Teoh YL, Tang H, Boudville I, Oostvogels LC, Suryakiran PV, Smolenov IV, Han HH, Bock HL. Safety and efficacy of human rotavirus vaccine during the first 2 years of life in Asian infants: randomised, double-blind, controlled study. Vaccine. 2009 Oct 9;27(43):5936-41. doi: 10.1016/j.vaccine.2009.07.098. Epub 2009 Aug 11. PMID 19679216
- [Background] Phua KB et al. Efficacy of rotavirus vaccine RIX4414 during the first 3 years of life: a randomised, double-blind, placebo-controlled study in infants from Hong Kong, Singapore and Taiwan. Abstract presented at the 10th International Rotavirus Symposium (IRS), Bangkok, Thailand, 19-21 Sep 2012.
- [Background] Phua KB et al. Human rotavirus vaccine RIX4414 (Rotarix™) is highly efficacious in Asian infants during the first three years of life. Abstract presented at the 13th Asian Pacific Congress of Pediatrics (APCP). Shanghai, China, 14-18 October 2009.
- [Background] Phua KB et al. Human rotavirus vaccine RIX4414 (Rotarix™) is highly efficacious in infants from Asia during the first two years of life. Abstract presented at the 13th International Congress on Infectious Diseases (ICID). Kuala Lumpur, Malaysia, 19-22 June 2008.
- [Background] Phua KB et al. Human rotavirus vaccine RIX4414 is highly efficacious in Asian infants during the third year of life. Abstract presented at the 27th Annual Meeting of the European Society for Paediatric Infectious Diseases (ESPID). Brussels, Belgium, 9-13 June 2009.
- [Derived] Lim FS, Phua KB, Lee BW, Quak SH, Teoh YL, Ramakrishnan G, Han HH, Van Der Meeren O, Jacquets JM, Bock HL. Safety and reactogenicity of DTPa-HBV-IPV/Hib and DTPa-IPV/I-Hib vaccines in a post-marketing surveillance setting. Southeast Asian J Trop Med Public Health. 2011 Jan;42(1):138-47. PMID 21323176
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 444563/028/029/030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 444563/028/029/030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 444563/028/029/030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 444563/028/029/030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 444563/028 are summarised with studies 444563/029, 444563/030, 107070, 107072, and 107076 on the GSK Clinical Study Register.
- Available data/document: Study Protocol: 444563/028/029/030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 444563/028/029/030 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register